CLINICAL TRIAL: NCT06515015
Title: Exploratory, Single-Group, Single-Center Clinical Study to Evaluate the Feasibility, Safety, and Efficacy of Single-use Endobronchial Silicon Spigots for the Treatment of Refractory Pneumothorax
Brief Title: Evaluation of the Feasibility, Safety, and Efficacy of Single-use Endobronchial Silicon Spigots for the Treatment of Refractory Pneumothorax
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Broncus Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-I-ESS-01
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Pneumothorax
Keywords: Pneumothorax; spigots; air leakage; bronchial occlusion
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Intervention Model Description: This study is a single-arm trial, intending to enroll 10 subjects. All subjects will be assigned to the treatment group to receive the study treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): All subjects will be assigned to the treatment group to receive the endobronchial silicon spigot treatment.
  Interventions: Device: Endobronchial Silicon Spigots

INTERVENTIONS:
Device: Endobronchial Silicon Spigots — The single-use endobronchial silicon spigot is injection-molded from implant-grade silicone and has a solid conical body. The endobronchial silicon spigot is used for the temporary occlusion of the target bronchus. It is delivered to the target bronchus through a bronchoscope using biopsy forceps, and the position of the blocker is adjusted to occlude the responsible bronchus leading to the pleural air leakage.

SUMMARY:
Study Objective: To evaluate the feasibility and safety of the disposable endobronchial silicon spigots for treating refractory pneumothorax and to preliminarily assess its efficacy, providing domestic experience for the development and clinical application of bronchial occlusion.

Study Population: Patients intended to receive selective bronchial occlusion technology for the treatment of refractory pneumothorax.

Sample Size: This study is a preliminary exploration of the application value of the disposable endobronchial silicon spigots occlusion technology in refractory pneumothorax. The sample size has not been strictly calculated, and it is expected to include 10 patients.

Study Design: This study is an exploratory, single-group, single-center clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be enrolled:

  1. Male or female, aged ≥18 years;
  2. Patients with various types of pneumothorax who still have persistent air leaks after continuous intercostal drainage for 7 days;
  3. After evaluation by the researcher, the subject is feasible for the bronchoscopic procedure of selective bronchial occlusion to treat refractory pneumothorax, and the responsible bronchus can be determined by the balloon detection;
  4. Voluntarily participate in this trial and sign an informed consent form.

Exclusion Criteria:

* Subjects with any of the following conditions cannot be selected:

  1. Allergic to silicone materials;
  2. Contraindications for bronchoscopy:

     * Myocardial infarction within the past month;
     * Active massive hemoptysis;
     * Platelet count <20×10^9/L;
     * Pregnancy;
     * Malignant arrhythmias, unstable angina, severe cardiopulmonary dysfunction, hypertensive crisis, severe pulmonary arterial hypertension, intracranial hypertension, acute cerebrovascular events, aortic dissection, aortic aneurysm, severe mental illness, and extreme systemic exhaustion, etc.
  3. Uncontrolled acute pulmonary infection or severe chronic infection at the intended occlusion lobes or segments;
  4. Obvious hemodynamic instability or unstable respiratory failure;
  5. The responsible bronchus cannot be determined by balloon detection;
  6. The researcher believes that the patient has other conditions that are not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Total Occlusion Success Rate | 7 days
  The percentage of subjects who are successfully* occluded after temporary embolization with endobronchial silicon spigots (including second occlusion) out of the total number of subjects receiving bronchial blocker treatment.

SECONDARY OUTCOMES:
First Occlusion Success Rate | 14 days
  The percentage of subjects who are successfully occluded after the first endobronchial silicon spigots treatment out of the total number of subjects receiving endobronchial silicon spigots treatment; if a second occlusion is received within 7 days after surgery, it is not counted as a first occlusion success.
First Occlusion Cure Rate | 14 days
  The percentage of subjects whose chest drainage tube completely stops leaking air within 14 days after the first endobronchial silicon spigots treatment out of the total number of subjects receiving endobronchial silicon spigots treatment; if a second occlusion is received within 14 days after surgery, it is not counted as a first occlusion cure.
Total Occlusion Cure Rate | 42 days
  The percentage of subjects whose chest drainage tube completely stops leaking air within 14 days after endobronchial silicon spigots treatment (including second occlusion) out of the total number of subjects receiving endobronchial silicon spigots treatment.
Chest Drainage Tube Removal Rate | 28 days
  The percentage of subjects who successfully remove the chest drainage tube within 28 days after endobronchial silicon spigots treatment (including second occlusion) out of the total number of subjects receiving endobronchial silicon spigots treatment.
Endobronchial spigots Removal Time | 30 days
  The time (in days) from successful placement of the endobronchial silicon spigots to successful removal of the endobronchial silicon spigots.
Technical Success Rate | 30 days
  The proportion of successful placements of the endobronchial silicon spigots into the responsible drainage bronchus out of the total number of operations.
Incidence of Treatment-Emergent Adverse Events | 30 days
  Record all adverse events during surgery and postoperative follow-up, assess the relatedness to the device itself and treatment, and calculate the incidence of device-related and surgical treatment-related adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Zeng, M.D, Principal Investigator — The Second Affiliated Hospital of Fujian Medical University
Locations (1):
- The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian, China